CLINICAL TRIAL: NCT06885008
Title: The Effects of Aerobic Exercise and Active Video Games as Adjuncts to Conventional Physiotherapy on Pain, Functional Capacity, and Balance in Knee Osteoarthritis
Brief Title: Effect of Video-based Game and Aerobic Exercise on Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Ass. Prof., Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/05
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis of Knee
Keywords: Knee Osteoarthritis; Video Games; Aerobic Exercise; Pain; Disabilitiy
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gaming (Experimental): The gaming group played active video games via Xbox kinect 3 days per week, addition to conventional physiotherapy for 8 weeks.
  Interventions: Other: Active video game; Other: Conventional treatment
- Aerobic (Experimental): The aerobic group engaged in cycling-based aerobic exercise (20 minutes per session) 3 days per week addition to conventional physiotherapy for 8 weeks.
  Interventions: Other: Aerobic exercise; Other: Conventional treatment
- Control (Experimental): The control group received only conventional physiotherapy and continued their daily activities.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Active video game — The participants played the video game using an Xbox 360 Kinect console connected to a 55-inch Full HD television. The video games were planned with the assistance of a physiotherapist, 3 days per week, with 8 repetitions during the first 4 weeks and 12 repetitions during the final 4 weeks. The warm-up and cool-down periods were designed and applicated.
  Arms: Gaming
Other: Aerobic exercise — Aerobic exercise training was performed on a stationary bike, 3 days per week, for 20 minutes per session. The intensity of the aerobic exercise was determined using the Karvonen method. For the first 4 weeks, the intensity was set at 30-50% of the maximum heart rate (MHR), corresponding to light intensity, and was then increased to 50-70% (moderate intensity) for the following 4 weeks. A pulse oximeter (ChoiceMMed, China) was used to monitor the target heart rate. During both the warm-up and cool-down phases of the aerobic exercise, participants performed hip abduction and adduction, hip-knee flexion, heel raises, and mini squats while standing for 3-5 minutes.
  Arms: Aerobic
Other: Conventional treatment — Convetional treatment included Hotpack, Transcutaneous Electrical Nerve Stimulation (TENS), and Ultrasound (US) modalities, were applied to the symptomatic knee(s) for a total duration of 30 minutes. Following this, the exercise program outlined below was performed with 3 sets of 10 repetitions each. The session lasted approximately 45 minutes.

SUMMARY:
This randomized controlled trial was conducted by the CONSORT guidelines for non-pharmacological treatments. Participants were randomly assigned to control, gaming, or aerobic groups using the closed-envelope randomization method. All groups received conventional physiotherapy for 8 weeks. In addition, the gaming group played active video games 3 days per week, while the aerobic group engaged in cycling-based aerobic exercise (20 minutes per session) 3 days per week. The control group received only conventional physiotherapy and continued their daily activities. Evaluations were performed by the same assessor at the baseline and after eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants, aged 30-65 years who were diagnosed with unilateral or bilateral osteoarthritis based on the clinical and radiological criteria of the American College of Rheumatology.
* The severity of osteoarthritis was classified as stage 2-3 according to the Kellgren-Lawrence grading system for gonarthrosis.
* Participants were required to be able to walk independently for at least 15 meters and to refrain from using non-steroidal anti-inflammatory drugs (NSAIDs) during the study period.

Exclusion Criteria:

* A history of lower extremity surgery within the past 6 months,
* The presence of neurological or systemic diseases,
* Other inflammatory joint diseases,
* Getting classic physiotherapy and rehabilitation within the past month,
* Intra-articular corticosteroid injections within the past 3 months,
* Severe joint deformities or movement restrictions,
* Severe visual impairments.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Knee disability | 8 weeks
  The WOMAC index was used to assess functional disability in patients with knee osteoarthritis. It consists of 24 items divided into three subcategories: pain severity, stiffness, and physical function. Each item is scored on a 5-point Likert scale ranging from 0 to 4. The total score is calculated as a percentage, with higher scores indicating increased pain and stiffness and reduced physical function.
Functional capacity | 8 weeks
  The 6MWT was used to measure patients' functional capacity. Two cones were placed 30 meters apart, and participants were instructed to walk as quickly as possible without running. The total distance walked in six minutes was recorded in (m) meters.
Functional Performance | 8 weeks
  The TUG test was administered to assess dynamic balance, walking speed, and functional performance. Participants were seated in a fixed chair without armrests, with their hips and knees positioned at a 90-degree angle. Upon the "START" command, they were instructed to stand up, walk three meters, turn around a designated cone, and return to the starting position. The total time (seconds) required to complete the task was recorded.
Balance | 8 weeks
  The modified Y-Balance test was used to assess dynamic balance. In this test, the maximum distances reached in the Anterior (A), Posteromedial (PM), and Posterolateral (PL) directions were recorded. The assessment was conducted using a specialized platform with Y-shape. Participants were instructed to position the foot being tested at the center of the platform while reaching as far as possible with the opposite foot in the A, PM, and PL directions. Measurements were taken bilaterally, ensuring that the participant's balance was maintained throughout the procedure. The test was repeated three times, and the average distances were recorded in (cm) centimeters.

SECONDARY OUTCOMES:
Limb strength | 8 weeks
  The strength of selected lower extremity muscles was measured using a hand-held dynamometer (HHD) (Model-01165, Lafayette Instrument®, Lafayette IN, USA), with results recorded in newtons. Quadriceps, hamstring, gluteus medius muscles strength were measured. Before strength measurements, each participant performed a familiarization trial. Three measurements were taken for each muscle group, and the average value was used for analysis. A 120-second rest period was provided between measurements,

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Usgu, Ass Prof, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Department of Physiotherapy and Rehabilitation, Şahinbey, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kong H, Wang XQ, Zhang XA. Exercise for Osteoarthritis: A Literature Review of Pathology and Mechanism. Front Aging Neurosci. 2022 May 3;14:854026. doi: 10.3389/fnagi.2022.854026. eCollection 2022. PMID 35592699
- [Background] Cicek A, Ozdincler AR, Tarakci E. Interactive video game-based approaches improve mobility and mood in older adults: A nonrandomized, controlled tri̇al. J Bodyw Mov Ther. 2020 Jul;24(3):252-259. doi: 10.1016/j.jbmt.2020.01.005. Epub 2020 Feb 6. PMID 32825997
- [Background] Oiestad BE, Aroen A, Rotterud JH, Osteras N, Jarstad E, Grotle M, Risberg MA. The efficacy of strength or aerobic exercise on quality of life and knee function in patients with knee osteoarthritis. A multi-arm randomized controlled trial with 1-year follow-up. BMC Musculoskelet Disord. 2023 Sep 8;24(1):714. doi: 10.1186/s12891-023-06831-x. PMID 37684597
- [Background] Lange B, Flynn S, Proffitt R, Chang CY, Rizzo AS. Development of an interactive game-based rehabilitation tool for dynamic balance training. Top Stroke Rehabil. 2010 Sep-Oct;17(5):345-52. doi: 10.1310/tsr1705-345. PMID 21131259